CLINICAL TRIAL: NCT00237198
Title: Study of Safety and Efficacy of Letrozole Monotherapy as Second-line Endocrine Therapy in Postmenopausal Patients With Advanced Breast Cancer Who Received Previous Anti-estrogen Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345F1203
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Postmenopausal Women With Advanced Breast Cancer
Keywords: Aromatase inhibitor; letrozole; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

ARMS (1):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole
  Other Names: FEM345

SUMMARY:
* Safety and efficacy of letrozole 2.5 mg/day monotherapy as second-line endocrine therapy in postmenopausal patients with advanced breast cancer who received previous anti-estrogen treatment
* To investigate changes in blood drug concentrations and blood hormone kinetics.
* To investigate gene polymorphisms of CYP2A6, an enzyme involved in the metabolism of letrozole

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically documented breast cancer
* Patients with progressive breast cancer (advanced breast cancer, locoregional recurrence not operative, or metastatic breast cancer)
* Patients with hormone receptor (ER and/or PgR) positive or both unknown.
* Postmenopausal patients between ages 20 and 79 years, inclusive
* Patients with a history of adjuvant therapy or advanced breast cancer treated with anti-estrogens
* Patients with documented measurable or evaluable lesions.
* Patients with sufficient organ function to evaluate the safety
* Patients whose performance status (PS) is 0～2

Exclusion Criteria:

* Patients with diffuse lymphangitis carcinomatosa of the lung or CNS involvement, liver metastasis occupying more than one third of the liver, or inflammatory breast cancer
* Patients with other concurrent or previous malignant disease (excluding contralateral breast cancer, in situ carcinoma of cervix uteri, and adequately treated basal or squamous cell carcinoma of the skin)
* Patients in whom one of the following is the sole manifestation of disease: hilar enlargement, pleural effusion and ascites
* Patients with only blastic bone metastases or a mixed blastic and lytic bone metastases at the same site and no other measurable or evaluable lesions
* Patients with serious current disease such as uncontrolled cardiac diseases and/or uncontrolled diabetes mellitus by any medications (including a historical serious cardiac disease)
* Patients with adrenal insufficiency (treated or untreated) or Cushing's syndrome
* Patients with any of the following previous treatments

  1. Chemotherapy for metastatic and/or locoregional recurrent disease
  2. Previous adjuvant endocrine therapy other than ovariectomy, anti-estrogen treatment, LH-RH analogues or radiation castration
  3. Previous first-line endocrine therapy (e.g., aromatase inhibitors and gastagens) for the treatment of metastatic and/or locoregional recurrent breast cancer other than anti-estrogen or LH-RH analogues treatment
  4. Patients who have not recovered from toxicity caused by previous therapy
  5. For patients on investigational drugs, adequate wash-out periods of at least 7 days in the case of topical investigational drugs and at least 30 days in the case of systemic
  6. Previous bisphosphonate therapy started within 6 months without any other measurable or evaluable lesions
  7. Patients who have not stopped treatment with other anti-estrogen or anti-cancer drugs (other than bisphosphonates) before starting the trial medication

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 20 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-03; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety during treatment | Until disease progression or appearance of unacceptable toxicity whichever comes first
Response Rate during treatment | Until disease progression or appearance of unacceptable toxicity whichever comes first

SECONDARY OUTCOMES:
Clinical Benefit Rate during treatment | Until disease progression or appearance of unacceptable toxicity whichever comes first
Duration of response | from the first date of response confirmed and the last date of response confirmed
Time to progression | from the first date of response confirmed and the last date of response confirmed
Time to treatment failure | from the date of study initiation and the date of disease progression confirmed or discontinuation other than disease progression
Plasma drug concentration from baseline, every 4 weeks until 28 weeks, at 40 weeks and at 52 weeks | Baseline, 52 weeks
Plasma estrogens level | baseline, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Japan (21):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, kooriyama, Fukushima
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Niigata, Niigata
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Cyuo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo